CLINICAL TRIAL: NCT01018082
Title: Longitudinal Study of Neurologic, Cognitive, and Radiologic Outcomes in PHACE Syndrome
Brief Title: Longitudinal Study of Neurologic, Cognitive, and Radiologic Outcomes of PHACE Syndrome
Acronym: PHACE
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Beth A Drolet, MD, Professor and Vice Chairman of Pediatric Dermatology, Medical College of Wisconsin
Other Study IDs: CHW09/140, GC 942
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: PHACE Syndrome
MeSH Terms: conditions — Aortic Aneurysm, Giant Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall goal of this 2-year pilot project is to utilize interdisciplinary strategies to determine the prevalence and type of neurodevelopmental impairment in PHACE syndrome, a rare vascular syndrome, and to rapidly translate discovery into clinical care guidelines that will identify at risk infants so early intervention can be initiated. Infantile hemangioma is the most common benign tumor of infancy, with an incidence estimated between 4-5%. A subgroup of patients with infantile hemangiomas exhibits additional associated structural anomalies of the brain, cerebral vasculature, eyes, aorta, heart, and chest wall in the rare neurocutaneous disorder called PHACE syndrome (OMIM 606519). PHACE refers to Posterior fossa anomalies, Hemangioma, Arterial lesions, Cardiac abnormalities/aortic coarctation, and abnormalities of the Eye. Affected children have multi-organ involvement, and an increasing number of cerebral, cerebellar, and cerebrovascular anomalies are being described; however, the significance of these neuroradiologic findings is not known. As the investigators' neonates with hemangiomas have grown into young children, neurodevelopmental impairment has become more evident, even among patients without MRI evidence of stroke or structural brain anomalies. Some infants develop progressive cerebral arterial disease leading to a moyamoya-like vasculopathy and ischemic stroke. An interdisciplinary research project studying brain and cerebral vascular imaging in concert with neurological, psychological, behavioral, neurodevelopmental, and quality of life outcome measures has never been conducted. Diagnostic and management guidelines are also lacking. The investigators' long-term goal is to develop medical and/or surgical therapeutic interventions that improve the overall health of children with PHACE syndrome. This novel project constitutes the first study of the most devastating feature of PHACE syndrome: the neurodevelopmental sequelae.

DETAILED DESCRIPTION:
Aim 1) Establish a cohort of 30 well-characterized patients with PHACE syndrome and enhance existing tissue and DNA banks to facilitate future investigation.

We will use rigorous phenotyping strategies to establish a cohort of 30 patients with PHACE syndrome 4-6 years of age, and collect neuroimaging studies and patient tissue and DNA samples to enhance an existing tissue repository to facilitate future studies, such as validation of biomarkers.

Aim 2) Determine the prevalence and describe the spectrum of neurodevelopmental impairment in a cohort of patients 4-6 years of age with PHACE syndrome.

Given the multiple risk factors for neurodevelopmental deficits in PHACE patients, we propose a comprehensive assessment of a cohort of patients 4-6 years of age, this age range represents a critical period, as it is the time that most children enter the formal educational system and it allows for a more thorough evaluation of neurodevelopmental skills. Upon completion of this 2-year study we expect to have immediate impact on clinical care by identifying specific deficits in this cohort. Once identified and quantified, we will publish the data with clinical guidelines for patient management including age and frequency of neuroimaging, frequency of neurologic evaluation, and age and utility of neurodevelopmental assessment. We anticipate that these guidelines will identify at risk infants and early intervention can be initiated, resulting in improved functional outcomes. In addition, this data will provide a cost-effective functional outcome methodology that can be used for clinical trials and to validate biomarkers identified in this pilot study.

Aim 3) Identify potential clinical, molecular, biochemical, and imaging biomarkers aimed at early detection and risk stratification of cerebrovasculopathy and neurodevelopmental impairment.

We hypothesize that certain risk factors including, but not limited to, genotype, hemangioma size, hemangioma location, cerebral anomalies, cerebellar anomalies, and cerebrovascular anomalies predispose patients to progressive vasculopathy. We will determine risk factors and identify biomarkers for progressive cerebrovascular disease. Based on this information we will establish guidelines for serial and diagnostic cerebrovascular imaging and develop a method of risk-stratification that will allow for early clinical prediction and intervention of long-term neurodevelopmental prognosis. Specific Aims

ELIGIBILITY:
Inclusion Criteria:

1. Fulfills definite or possible PHACE syndrome diagnostic criteria, per consensus statement November 2008;
2. Child is between 4-6 years of age; and
3. Parents able and willing to travel to our center (Medical College of Wisconsin) for evaluations.

Exclusion Criteria:

1. Patients with known genetic disorders in addition to PHACE syndrome;
2. Patients unable to undergo adequate MR imaging due to pacemaker or other MRI-incompatible implant(s); or
3. Non-English and non-Spanish speaking patients will be excluded due to interpreter-related inconsistencies in neurocognitive testing. Clinical Evaluation: A standardized electronic data collection form will be designed. Demographic data, clinical -

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between the ages of 4-6 years who fulfill the diagnostic criteria for PHACE syndrome will be contacted for enrollment.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Establish a cohort of 30 patients 4-6 years of age, define the functional and neurodevelopmental outcome of PHACE syndrome, and identify potential biomarkers that predict progressive vasculopathy, ischemic stroke, and neurodevelopmental impairment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Beth Drolet, MD, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Childrens Hospital of Wisconsin, Milwaukee, Wisconsin, United States